CLINICAL TRIAL: NCT00584909
Title: A Phase II Study of Paclitaxel and Carboplatin in Patients With Intermediate-Risk Adenocarcinoma of the Endometrium
Brief Title: A Phase II Study of Paclitaxel and Carboplatin in Patients With an Elevated-Risk Cancer of the Uterus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, J. Michael Straughn, MD, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F060328016 (UAB 0604); UAB 0604 (Other: UAB Department study number)
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Results first posted 2012-03-29 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Uterine Cancer
MeSH Terms: conditions — Uterine Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open Label (Experimental)
  Interventions: Drug: Paclitaxel and carboplatin combination

INTERVENTIONS:
Drug: Paclitaxel and carboplatin combination — Paclitaxel will be administered at an appropriate dose (175 mg/m2) as a 3-hour continuous IV infusion every 21 days. Carboplatin will be administered at an appropriate dose utilizing the Calvert formula for determining the area under the curve (AUC) based on the patient's glomerular filtration rate (GFR).

SUMMARY:
The main purpose of this study us to determine the best treatment for patients with endometrial cancer who are at an elevated risk for recurrence.

DETAILED DESCRIPTION:
Endometrial cancer is the most common gynecologic malignancy in the United States with 40,880 new cases diagnosed and 7,310 deaths attributable to this malignancy expected in 2005. The majority of patients diagnosed with endometrial cancer have early stage disease that is amenable to treatment with hysterectomy and bilateral salpingo-oophorectomy with excellent clinical outcomes. Surgical staging has improved accuracy over clinical staging for defining a low-risk population of patients who have favorable long-term outcomes with surgery alone. However, approximately 10-15% of patients with surgical stage I endometrial carcinoma (confined to the uterus) will have invasion to the outer one-half of the myometrium (stage IC) and a moderately to poorly differentiated tumor (grade 2 or 3). These patients are at a higher risk for recurrence (approximately 20-25% recurrence rate over 5 years). This patient population has been historically considered at "intermediate-risk" for recurrence because they are at lower risk than patient with disease spread beyond the uterus, but higher risk than patients with a grade 1 tumor or minimally invasive (Stage IA or IB). The optimal mode of postoperative management for this population of patients has yet to be defined.

Historically, radiation therapy has been used in some form in patients diagnosed with intermediate-risk endometrial cancer. Two randomized trials published in the last 5 years have evaluated the use of adjuvant radiation therapy in patients with intermediate-risk endometrial adenocarcinoma. the Gynecologic Oncology Group (GOG) studied the use of adjuvant whole pelvic radiation (WPRT) versus no adjuvant therapy (NAT) in patients with stage IB, IC, and II (occult)endometrial adenocarcinoma. In a study of 392 patients, the use of WPRT had a substantial impact on local recurrences (18 in NAT versus 3 in WPRT), but had no impact on the risk of distant recurrence (18 NAT versus 11 in WPRT). Because of the lack of distant control, the use of WPRT did not impact overall survival (estimated 4 year survival 86% in NAT versus 92% in WPRT, p=0.557). The PORTEC trial randomized patients with intermediate-risk Stage I endometrial carcinoma to WPRT versus NAT. Of note, patients in this trial were not surgically staged. Of 714 patients with a median follow-up of 52 months,local recurrence rates were 4% in the WPRT group versus 14% in the control group (p<0.001). The use of WPRT did not impact 5-year overall survival (81% WPRT versus 85% NAT). Furthermore, some clinicians have advocated observation after surgical staging with radiation therapy reserved for those patients who recur locally. Several reports have reported salvage rates of 50-66% for patients with local recurrences. Given that approximately 20-25% patients in this population will recur locally, many clinicians prefer to use local radiation therapy as salvage therapy, thus sparing the majority of patients the potential long-term effects of pelvic radiation therapy. Given that radiation therapy does not affect distant metastasis and carries significant long-term morbidity, other therapies are necessary to improve disease-free survival in this setting. Adjuvant systemic chemotherapy is one potential option for these patients since it may sterilize both local and distant metastases. The use of adjuvant chemotherapy may be more desirable than radiation therapy because most side effects of chemotherapy are short-term and subside once therapy is completed or discontinued.

Multiple chemotherapeutic agents including cisplatin, doxorubicin HCL, paclitaxel, carboplatin, and oral etoposide have been studied for patients with advanced or recurrent endometrial cancer. A phase III study by the Gynecologic Oncology Group (GOG) compared doxorubicin with and without cisplatin (GOG 107) for patients with advanced or recurrent endometrial cancer. A higher response rate (42% vs. 25%) was noted for combination therapy and has been considered by many to be the standard chemotherapy regimen for treatment of patients with advanced endometrial cancer. Paclitaxel has also been studied as a single agent and in combination with platinum compounds in this setting. A phase II study that combined paclitaxel 175 mg/m2 as a 3-hour infusion with cisplatin 75 mg/m2 reported a 67% response rate. There were seven complete responses and nine partial responses with an 18-month median overall survival. An additional phase II study evaluated the efficacy of combining paclitaxel and carboplatin in both primary and recurrent non-papillary and papillary tumors following radiation therapy. the response rate was 78% in patients with primary advanced non-papillary tumors with a median disease-free survival of 23 months, with the median overall survival of 15 months. Currently, many clinicians are using a combination of paclitaxel, doxorubicin, and cisplatin (TAP), based on a phase III GOG study that demonstrated not only a significantly higher response rate (57% vs. 33%) over the combination of doxorubicin and cisplatin (AP), but also a survival advantage (median, 15.3 vs. 12.3 months; P=.037). Significantly more neurotoxicity was experienced by patients in the TAP arm. Currently, the GOG is evaluating the TAP combination versus the more tolerable regimen of paclitaxel and carboplatin in a phase III setting.

The combination of paclitaxel and carboplatin is considered the standard of care for both high-risk early stage ovarian cancer and advanced ovarian cancer. The safety of this combination is well established in a number of phase III trials and currently is used in the primary setting for patients with ovarian cancer and advanced endometrial cancer. Although this combination is considered active in endometrial carcinoma, there is a paucity of data regarding the use of adjuvant chemotherapy in the setting of intermediate-risk endometrial adenocarcinoma. Accordingly, this phase II study will evaluate the combination of paclitaxel and carboplatin as adjuvant therapy for patients with early stage adenocarcinoma of the endometrium at elevated-risk for recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a elevated risk, surgical stage II, stage IC, grade 2 or 3 adenocarcinoma of the endometrium.
* Patients must have undergone, a total abdominal hysterectomy, bilateral salpingo-oophorectomy, peritoneal washings, and a pelvic and para-aortic lymphadenectomy.
* Patients must have adequate organ function defined as:

  1. Platelets >/= 100,000/µ
  2. Granulocytes (ANC)>/= 1,500/µl
  3. Creatinine</= 1.6 mg/dl
  4. SGOT (AST) </= 3x upper limits of normal
  5. Bilirubin within institutional normal limits
* Patients must have adequate performance status (ECOG performance status 0-2 or Karnofsky Performance Status >40)
* Patients must be age 19 or greater and have signed informed consent.

Exclusion Criteria:

* Patients with history of other malignancies within 5 years (except non- melanoma skin cancer or carcinoma-in-situ of the cervix) are ineligible.
* Patients with high-risk histologic subtypes of endometrial cancer such as papillary serous or clear cell histology are ineligible.
* Patients with histologic evidence of uterine sarcoma, including leiomyosarcoma, carcinosarcoma, endometrial stromal sarcoma, and adenosarcoma are ineligible.
* Patients who have received past pelvic radiotherapy are ineligible.
* Patients receiving any other investigational agents are ineligible.
* Patients with known hypersensitivity to paclitaxel and/or carboplatin are ineligible.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-03; Primary Completion 2010-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M. Straughn, MD, Principal Investigator — Assistant Professor, Dept of OB/Gyn, Division of GYN Oncology
Locations (1):
- UAB Women's and Infant Center, 1700 6th Avenue South, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Paclitaxel + Carboplatin: Patients are administered 175 mg/m2 paclitaxel and carboplatin (dose based upon the Calvert formula for determining the area under the curve based on the patient's glomerular filtration rate). Drugs will be administered by intravenous infusion every 21 days for 6 cycles.
Period: Overall Study
Arm/Group | Paclitaxel + Carboplatin
Started | 13
Completed | 9
Not Completed | 4
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Arm/Group | Paclitaxel + Carboplatin
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival
Description: Number of months of survival with no evidence of disease
Time Frame: 4 years - Median follow up time of 45.3 months
Measure: Median (Full Range); unit: months
Arm/Group | Paclitaxel + Carboplatin
Number analyzed (Participants) | 9
months | 50.5 [35.5 to 55.9]

2. Secondary Outcome: Toxicity
Description: Toxicity secondary to paclitaxel and carboplatin based upon the NCI common toxicity criteria version
Time Frame: 4 years
Measure: Number; unit: participants
Arm/Group | Paclitaxel + Carboplatin
Number analyzed (Participants) | 9
participants | 9

ADVERSE EVENTS:
Arm/Group | Paclitaxel + Carboplatin
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 9/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel + Carboplatin (N=9)
Neutropenia (Immune system disorders) | 6 (12)
Neuropathy (Nervous system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Gastrointestinal (Gastrointestinal disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early due to slow accrual. 4 patients withdrew from the study due to side-effects from the treatment. All 9 patients were evaluable for toxicity and PFS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes